CLINICAL TRIAL: NCT00469521
Title: Pilot Study Evaluation of 2 Artificial Tears. Evaluation of TBUT, Tear Meniscus Height and Tear Thickness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 5304
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Tear Film Thickness

INTERVENTIONS:
Drug: Refresh Tears, 9582X

SUMMARY:
To determine baseline tear thickness and improvement immediately post installation of two artificial tear solutions:(9582X) and Allergan Refresh Tears.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy volunteers 18 years or older
2. Males or females
3. Any race or ethnic background

Exclusion Criteria:

1. Corneal refractive surgery within 6 months of this study.
2. Contact lens use on day of examination.
3. Corneal ectasia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Helga Sandoval, MS, MD, Principal Investigator — Magill Research Center Institute MUSC
Locations (1):
- Magill Research Center Institute MUSC, Charleston, South Carolina, United States